CLINICAL TRIAL: NCT04944836
Title: Sex Hormone Supplementation and Rotator Cuff Repair: A Preliminary Randomized Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Peter Chalmers, Associate Professor, Department of Orthopaedic Surgery, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCRHRT
Record Dates: First submitted 2021-06-08; First posted 2021-06-30 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): All patients will receive non-labeled pills identical in appearance from our pharmacy, to be taking once every other day. In the control group, these will be placebo. These will be taken every other day for seven months beginning four week prior to surgery and extending for six months after surgery.
  Interventions: Procedure: Rotator Cuff Repair
- Clomiphene (Experimental): All patients will receive non-labeled pills identical in appearance from our pharmacy, to be taking once every other day. In the study group, these will contain 50 mg of clomiphene citrate. These will be taken every other day for seven months beginning four week prior to surgery and extending for six months after surgery.
  Interventions: Drug: Clomiphene Citrate; Procedure: Rotator Cuff Repair

INTERVENTIONS:
Drug: Clomiphene Citrate — All patients will receive non-labeled pills identical in appearance from our pharmacy, to be taking once every other day. In the study group, these will contain 50 mg of clomiphene citrate. In the control group, these will be placebo. These will be taken every other day for seven months beginning four weeks prior to surgery and extending for six months after surgery. After enrollment patients will be randomized. Patient will be assigned to the 2 groups using a permuted block randomization scheme with blocks of size 2, 4, and 6. Prior to initiation of the study opaque sealed envelopes will be prepared and thoroughly shuffled and then used sequentially during the study. These randomization assignments will be available to the pharmacy in a web-based format or by cards in sealed envelopes. A nonparticipant in the study (the pharmacy at our institution) will administer this process.
  Arms: Clomiphene
Procedure: Rotator Cuff Repair — The operative protocol will be standardized in all patients. Both the operative protocol and post-operative rehabilitation protocol will be per our standard of care, without alteration. An arthroscopic approach will be used. In all cases a double-row rotator cuff repair using triple-loaded anchor(s) on the medial row will be used. Post-operatively all patients will be placed in a sling for six weeks. Active range of motion exercises will begin at six weeks post-operatively and strengthening will be delayed until 12 weeks post-operatively. In all phases of care our peri-operative and post-operative protocol for study patients will be similar to our current clinical practice to ensure generalizability.

SUMMARY:
Shoulder tendon tears are a common cause of shoulder pain and disability and after surgery the repaired tendon often does not heal. In this pilot study, men with low sex hormone levels will be randomly assigned to receive sex hormone therapy or placebo pills while healing from tendon repair surgery in their shoulder. Sex hormone therapy increases sex hormone levels, and the investigators will test whether these increased sex hormone levels show promise in improving tendon healing and patient shoulder function and pain.

DETAILED DESCRIPTION:
The rotator cuff is a system of tendons in the shoulder that stabilize the ball within the socket. These tendons frequently tear with age, which causes pain, weakness, and dysfunction in the shoulder. While these tears can be surgically repaired, they do not always heal. Our data suggest that deficiency of testosterone and estrogen can contribute to both tearing of the rotator cuff and failure of healing after rotator cuff repair. Testosterone can be converted into estrogen in the body through the aromatase enzyme, which is in both tendons and bones, as well as other tissues. Both testosterone and estrogen can improve bone quality. While testosterone is frequently prescribed for testosterone deficiency, when it is given your body no longer has the drive to make testosterone. So when the treatment is withdrawn testosterone levels can go very low until feedback mechanisms in the body motivate it to make more. As a result, testosterone is not usually given temporarily. For temporary treatment clomiphene avoids this issue. Clomiphene works at the feedback mechanisms within the body to trick the body into thinking testosterone and estrogen levels are low and thus to motivate it to make more testosterone and estrogen. However, clomiphene can only be given continuously to men, because women's estrogen levels regularly cycle up and down on a monthly basis and clomiphene interferes with this cycle. The purpose of this study is to determine whether clomiphene treatment decreases pain and improves function, increases tendon healing, and improves bone quality with rotator cuff repair in men. We hypothesize that clomiphene treatment will decrease pain and improve function, improve tendon healing, and improve bone quality with rotator cuff repair in men. This is a placebo-controlled study, so a control group of patients will received placebo pills, i.e. "sugar pills", instead of clomiphene. This is a randomized study, so patients enrolled in the study will be randomly assigned to the clomiphene group or the placebo group. This is a blinded study, so both the patients enrolled in the will not know whether they are in the clomiphene or the control group. This is a double-blinded study, so the doctors performing the surgeries and the study will not know whether each specific patient is in the clomiphene or the control group. Study participants will first start the clomiphene treatment one month before surgery and will continue the treatment for six months after surgery. Both before surgery and six months after surgery, study participants will fill out study questionnaires about shoulder pain and function. Both before surgery and six months after surgery, study participants will undergo an magnetic resonance imaging study to examine the rotator cuff tendons as well as the bone quality within the shoulder. The magnetic resonance imaging study after surgery is provided free to study participants. Study participants will be compensated for completing the study. These results are important because may lead to a better understanding of the problem, more effective treatment, and improved clinical outcomes for future patients.

ELIGIBILITY:
Inclusion Criteria

1. A plan for a primary rotator cuff repair
2. Male sex
3. >1 cm tear width, full thickness supraspinatus/infraspinatus tear

Exclusion Criteria

1. Active infection
2. Pre-operative testosterone supplementation
3. Known diagnosis of secondary testicular failure or testosterone deficiency
4. Medically unfit for operative intervention
5. Revision surgery
6. Unwillingness to participate in the study, including post-operative imaging
7. Inability to read or comprehend written instructions
8. Prisoner
9. Concomitant patch augmentation or tendon-transfer
10. Untreated prostate cancer
11. Liver disease
12. Pituitary or hypothalamic dysfunction

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) tendon healing Post-op | To be collected at 6 months (±4 weeks) post-operatively.
  MRI scans will be assessed by observers blinded to the patient's allocation. For each patient, the post-operative MRI will be categorized as either "healed" or "non-healed". On post-operative MRI only those patients without tendon defects will be considered to be healed. This will be the primary outcome of the study. The investigators have previously demonstrated this measurement to be reliable.

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Score Pre-op | To be collected within six months pre-operatively.
  The ASES score is a patient survey that creates a score on a 100 point scale incorporating questions regarding shoulder pain and shoulder function. This survey contains 11 questions and takes ~3 minutes to complete. Higher scores indicate a better outcome.
American Shoulder and Elbow Surgeons (ASES) Score 6 weeks | To be collected at six weeks (±2 weeks) post-operatively.
  The ASES score is a patient survey that creates a score on a 100 point scale incorporating questions regarding shoulder pain and shoulder function. This survey contains 11 questions and takes ~3 minutes to complete. Higher scores indicate a better outcome.
American Shoulder and Elbow Surgeons (ASES) Score 12 weeks | To be collected at 12 weeks (±2 weeks) post-operatively.
  The ASES score is a patient survey that creates a score on a 100 point scale incorporating questions regarding shoulder pain and shoulder function. This survey contains 11 questions and takes ~3 minutes to complete. Higher scores indicate a better outcome.
American Shoulder and Elbow Surgeons (ASES) Score 6 months | To be collected at 6 months (±4 weeks) post-operatively.
  The ASES score is a patient survey that creates a score on a 100 point scale incorporating questions regarding shoulder pain and shoulder function. This survey contains 11 questions and takes ~3 minutes to complete. Higher scores indicate a better outcome.
Simple Shoulder Test (SST) Score Pre-op | To be collected within six months pre-operatively.
  The SST score is a patient survey that creates a score on a 12 point scale incorporating questions regarding shoulder function. This survey contains 12 questions and takes ~3 minutes to complete. Higher scores indicate a better outcome.
Simple Shoulder Test (SST) Score 6 weeks | To be collected at six weeks (±2 weeks) post-operatively.
  The SST score is a patient survey that creates a score on a 12 point scale incorporating questions regarding shoulder function. This survey contains 12 questions and takes ~3 minutes to complete. Higher scores indicate a better outcome.
Simple Shoulder Test (SST) Score 12 weeks | To be collected at 12 weeks (±2 weeks) post-operatively.
  The SST score is a patient survey that creates a score on a 12 point scale incorporating questions regarding shoulder function. This survey contains 12 questions and takes ~3 minutes to complete. Higher scores indicate a better outcome.
Simple Shoulder Test (SST) Score 6 months | To be collected at 6 months (±4 weeks) post-operatively.
  The SST score is a patient survey that creates a score on a 12 point scale incorporating questions regarding shoulder function. This survey contains 12 questions and takes ~3 minutes to complete. Higher scores indicate a better outcome.
Visual Analogue Score (VAS) for pain Pre-op | To be collected within six months pre-operatively.
  The VAS pain score is a patient survey that creates a score on a 10 point scale incorporating a single question regarding shoulder pain. This survey takes <1 minute to complete. Lower scores indicate a better outcome.
Visual Analogue Score (VAS) for pain 6 weeks | To be collected at six weeks (±2 weeks) post-operatively.
  The VAS pain score is a patient survey that creates a score on a 10 point scale incorporating a single question regarding shoulder pain. This survey takes <1 minute to complete. Lower scores indicate a better outcome.
Visual Analogue Score (VAS) for pain 12 weeks | To be collected at 12 weeks (±2 weeks) post-operatively.
  The VAS pain score is a patient survey that creates a score on a 10 point scale incorporating a single question regarding shoulder pain. This survey takes <1 minute to complete. Lower scores indicate a better outcome.
Visual Analogue Score (VAS) for pain 6 months | To be collected at 6 months (±4 weeks) post-operatively.
  The VAS pain score is a patient survey that creates a score on a 10 point scale incorporating a single question regarding shoulder pain. This survey takes <1 minute to complete. Lower scores indicate a better outcome.
Magnetic Resonance Imaging (MRI) proximal humeral bone quality Pre-op | To be collected within six months pre-operatively.
  Both the pre-operative and post-operative MRI scans will include a ultra-short time-echo (UTE) coronal sequence. On the UTE sequence, maximum humeral cortical thickness will be measured orthogonal to the axis of the shaft five, ten, and fifteen cm distal to the top the head, as we have previously demonstrated this measurement to be accurate and reliable.
Magnetic Resonance Imaging (MRI) proximal humeral bone quality Post-op | To be collected at 6 months (±4 weeks) post-operatively.
  Both the pre-operative and post-operative MRI scans will include a ultra-short time-echo (UTE) coronal sequence. On the UTE sequence, maximum humeral cortical thickness will be measured orthogonal to the axis of the shaft five, ten, and fifteen cm distal to the top the head, as we have previously demonstrated this measurement to be accurate and reliable.
Strength Assessment Pre-op | To be collected within six months pre-operatively.
  Rotator cuff strength, as measured with a handheld dynamometer, will be measured. Abduction strength will be measured at 30 degrees of flexion, 30 degrees of abduction, neutral rotation, and full elbow extension. External rotation strength will be measured with the arm in adduction, neutral rotation, and 90 degrees of elbow flexion. These measures will be performed by a single research coordinator.
Strength Assessment 6 weeks | To be collected at six weeks (±2 weeks) post-operatively.
  Rotator cuff strength, as measured with a handheld dynamometer, will be measured. Abduction strength will be measured at 30 degrees of flexion, 30 degrees of abduction, neutral rotation, and full elbow extension. External rotation strength will be measured with the arm in adduction, neutral rotation, and 90 degrees of elbow flexion. These measures will be performed by a single research coordinator.
Strength Assessment 12 weeks | To be collected at 12 weeks (±2 weeks) post-operatively.
  Rotator cuff strength, as measured with a handheld dynamometer, will be measured. Abduction strength will be measured at 30 degrees of flexion, 30 degrees of abduction, neutral rotation, and full elbow extension. External rotation strength will be measured with the arm in adduction, neutral rotation, and 90 degrees of elbow flexion. These measures will be performed by a single research coordinator.
Strength Assessment 6 months | To be collected at 6 months (±4 weeks) post-operatively.
  Rotator cuff strength, as measured with a handheld dynamometer, will be measured. Abduction strength will be measured at 30 degrees of flexion, 30 degrees of abduction, neutral rotation, and full elbow extension. External rotation strength will be measured with the arm in adduction, neutral rotation, and 90 degrees of elbow flexion. These measures will be performed by a single research coordinator.
Range of motion Pre-op | To be collected within six months pre-operatively.
  Range of motion will be recorded. Research personnel experienced with the use of video will measure active abduction, active forward elevation, active internal rotation in adduction , and active external rotation in adduction. These will be measured sequentially during a single continuous video, first with the video viewing from anteriorly while the subject abducts while standing against a wall, then while viewing from laterally while the subject elevates while standing adjacent to a wall, then while viewing from posteriorly while the subject internally rotates in adduction, and then while viewing from superiorly while the subject externally rotates while sitting in a chair. This protocol has been previously used in many publications. These videos will be saved using subject numbers and then evaluated using a digital protractor by a third-party observer.
Range of motion 6 weeks | To be collected at six weeks (±2 weeks) post-operatively.
  Range of motion will be recorded. Research personnel experienced with the use of video will measure active abduction, active forward elevation, active internal rotation in adduction , and active external rotation in adduction. These will be measured sequentially during a single continuous video, first with the video viewing from anteriorly while the subject abducts while standing against a wall, then while viewing from laterally while the subject elevates while standing adjacent to a wall, then while viewing from posteriorly while the subject internally rotates in adduction, and then while viewing from superiorly while the subject externally rotates while sitting in a chair. This protocol has been previously used in many publications. These videos will be saved using subject numbers and then evaluated using a digital protractor by a third-party observer.
Range of motion 12 weeks | To be collected at 12 weeks (±2 weeks) post-operatively.
  Range of motion will be recorded. Research personnel experienced with the use of video will measure active abduction, active forward elevation, active internal rotation in adduction , and active external rotation in adduction. These will be measured sequentially during a single continuous video, first with the video viewing from anteriorly while the subject abducts while standing against a wall, then while viewing from laterally while the subject elevates while standing adjacent to a wall, then while viewing from posteriorly while the subject internally rotates in adduction, and then while viewing from superiorly while the subject externally rotates while sitting in a chair. This protocol has been previously used in many publications. These videos will be saved using subject numbers and then evaluated using a digital protractor by a third-party observer.
Range of motion 6 months | To be collected at 6 months (±4 weeks) post-operatively.
  Range of motion will be recorded. Research personnel experienced with the use of video will measure active abduction, active forward elevation, active internal rotation in adduction , and active external rotation in adduction. These will be measured sequentially during a single continuous video, first with the video viewing from anteriorly while the subject abducts while standing against a wall, then while viewing from laterally while the subject elevates while standing adjacent to a wall, then while viewing from posteriorly while the subject internally rotates in adduction, and then while viewing from superiorly while the subject externally rotates while sitting in a chair. This protocol has been previously used in many publications. These videos will be saved using subject numbers and then evaluated using a digital protractor by a third-party observer.

OTHER OUTCOMES:
Serum Hormone Measurement Surgery | To be collected at the time of surgery.
  Blood will be drawn and the following serum laboratory values will be collected: testosterone, bio-available testosterone, estradiol, all of which are reported in ng/dL.
Luteinizing Hormone Measurement Surgery | To be collected at the time of surgery.
  Blood will be drawn and serum luteinizing hormone values will be collected. These are reported in IU/L.
Serum Hormone Measurement 12 weeks | To be collected at 12 weeks (±2 weeks) post-operatively.
  Blood will be drawn and the following serum laboratory values will be collected: testosterone, bio-available testosterone, and estradiol, all of which are reported in ng/dL.
Luteinizing Hormone Measurement 12 weeks | To be collected at 12 weeks (±2 weeks) post-operatively.
  Blood will be drawn and serum luteinizing hormone values will be collected. These are reported in IU/L.
Pill Count Surgery | To be collected at the time of surgery.
  Subjects will be asked how many pills they have taken to determine patient compliance. Deviations from protocol will be recorded.
Pill Count 6 weeks | To be collected at six weeks (±2 weeks) post-operatively.
  Subjects will be asked how many pills they have taken to determine patient compliance. Deviations from protocol will be recorded.
Pill Count 12 weeks | To be collected at 12 weeks (±2 weeks) post-operatively.
  Subjects will be asked how many pills they have taken to determine patient compliance. Deviations from protocol will be recorded.
Pill Count 6 months | To be collected at 6 months (±4 weeks) post-operatively.
  Subjects will be asked how many pills they have taken to determine patient compliance. Deviations from protocol will be recorded.
Averse Event Assessment Surgery | To be collected at the time of surgery.
  At each visit patients will be queried regarding adverse events. Patients will asked about the following specific adverse events side effects: anxiety, decreased energy/fatigue, mood instability, difficulty sleeping, decreased libido, visual changes, bleeding, infection, complications from anesthesia, the need for further surgery. In addition, any post-operative injections will be recorded.
Averse Event Assessment 6 weeks | To be collected at six weeks (±2 weeks) post-operatively.
  At each visit patients will be queried regarding adverse events. Patients will asked about the following specific adverse events side effects: anxiety, decreased energy/fatigue, mood instability, difficulty sleeping, decreased libido, visual changes, bleeding, infection, complications from anesthesia, the need for further surgery. In addition, any post-operative injections will be recorded.
Averse Event Assessment 12 weeks | To be collected at 12 weeks (±2 weeks) post-operatively.
  At each visit patients will be queried regarding adverse events. Patients will asked about the following specific adverse events side effects: anxiety, decreased energy/fatigue, mood instability, difficulty sleeping, decreased libido, visual changes, bleeding, infection, complications from anesthesia, the need for further surgery. In addition, any post-operative injections will be recorded.
Averse Event Assessment 6 months | To be collected at 6 months (±4 weeks) post-operatively.
  At each visit patients will be queried regarding adverse events. Patients will asked about the following specific adverse events side effects: anxiety, decreased energy/fatigue, mood instability, difficulty sleeping, decreased libido, visual changes, bleeding, infection, complications from anesthesia, the need for further surgery. In addition, any post-operative injections will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No